CLINICAL TRIAL: NCT02206516
Title: Using Combined Neuroimaging Techniques and Clinical Measures to Assess Feasibility of tDCS as an Intervention in Adult ADD.
Brief Title: Feasibility of Transcranial Direct Current Stimulation (tDCS) in the Treatment of Adult Attention Deficit Disorder (ADD).
Acronym: BMST
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: ElMindA Ltd (Industry); Brainsway (Industry); Ornim Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0214-14
Record Dates: First submitted 2014-07-28; First posted 2014-08-01 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Adult Attention Deficit Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients (Experimental): Stimulation using tDCS will be administered daily, 5 days a week for 4 weeks. each session will last 22 minutes during which the anode electrode will be positioned over the right Inferior Frontal Gyrus (IFG) and the Katode electrode over the right Orbito Frontal Gyrus (OFG).
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation
  Other Names: neuroConn GmbH, Germany

SUMMARY:
This study aims at combining imaging techniques and clinical evaluations to assess clinical change as well as brain changes that occur as a result of brain stimulation in adult attention deficit disorder.

DETAILED DESCRIPTION:
This study will use clinical measures and cognitive tasks covering 3 different functional domains during functional magnetic resonance imaging (fMRI), ElectroEncephaloGram (EEG) and Ultrasound tagged near infrared spectroscopy (UT-NIRS), to assess functional brain changes as a result of a treatment protocol with Transcaranial direct current stimulation (tDCS) in adults suffering from attention deficit disorder (ADD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the ages of 18-65(male and female)
2. Diagnosed as suffering from Attention-Deficit Hyperactivity Disorder according to the DSM IV
3. Patients taking medication for ADHD will give their consent to stop those medication 48 before entering the study and throughout the daily treatments.
4. Gave informed consent for participation in the study
5. If referred by the treating psychiatrist, he or she approves of the subjects participation in the study

Exclusion Criteria:

1. Suffering from other diagnosis on axis 1
2. History of drug or alcohol abuse during the last year
3. Inability to achieve satisfying level of communication with the subject

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy will be examined by the change in the CAARS questionnaire from the baseline visit to the determination visit in the treatment group compared to the control group. | 6 weeks

SECONDARY OUTCOMES:
changes in functional activity after 4 weeks of tDCS treatment during response inhibition | 6 weeks
  ROI analysis of right Inferior frontal cortex will be measured during response inhibition in the Go/Nogo task at the end of the 4 weeks of treatment and will be compared to baseline measures.

CONTACTS AND LOCATIONS:
Overall Officials: Talma Hendler, MD, PhD, Principal Investigator — TASMC
Locations (1):
- TASMC, Tel Aviv, Israel